CLINICAL TRIAL: NCT06149780
Title: Efficacy and Safety of the Fractionated 1927-nm Non Ablative Thulium Laser in Treating Post Inflammatory Hyperpigmentation in Skin Phototypes IV-VI
Brief Title: Fractionated 1927-nm Non Ablative Thulium Laser in Treating Post Inflammatory Hyperpigmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Tasneem Mohammad, Staff Physician, Department of Dermatology, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16268
Record Dates: First submitted 2023-10-24; First posted 2023-11-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fractional laser patients treated with laser (Experimental): Laser with topical steroid and laser with vehicle.
  Interventions: Device: Patients treated with laser

INTERVENTIONS:
Device: Patients treated with laser — Patients treated with laser with topical steroid Patients treated with laser with vehicle

SUMMARY:
To study the effect of fractionated 1927-nm non ablative thulium laser in reduction of post inflammatory hyperpigmentation (PIH) using a validated and reproducible model for studying PIH.

* Determine if there is aa reduction in PIH in patients treated with three (3) monthly sessions of fractionated 1927-nm non ablative thulium laser
* Determine if there is efficacy of post-procedure clobetasol propionate 0.05% ointment in the management of PIH
* Determine the histological and molecular changes that occur with laser and laser plus topical steroid treatment compared to untreated skin

DETAILED DESCRIPTION:
The design of the study consists of a total of six visits including one initial screening visit within 107-127 days depending on the scheduling of your screening and subsequent visits. Assessments such as visual examination, photography, Investigatory Global Assessment (IGA) of pigmentation and erythema; Colorimetry; and Diffuse Reflectance Spectroscopy of the intended treatment area will be conducted at Visits 1-5. Optional biopsies will be taken at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 and older
* Patient with skin phototypes IV-VI
* Patient able to understand requirements of the study and risks involved
* Patient able to sign a consent form
* Patient to have discontinued all oral medications used to treat pigmentary abnormalities and all topical medications, except for sunscreen, used to treat pigmentary abnormalities on the buttocks one month prior to treatment

Exclusion Criteria:

* A patient who has skin dyspigmentation, birth marks, tattoos, or other skin findings at baseline on either buttock that may obscure study results
* A patient who is lactating, pregnant, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Degree of Pigmentation in all 5 subjects | Visit 1 (Day 0) through Visit 5 (Day 112 ±5)
  Measured clinical with IGA objectively with colometry

SECONDARY OUTCOMES:
Immunohistochemical changes in pigmentation in all 5 subjects | Visit 2 (Day 28±5) and Visit 5 (Day 112 ±5)
  Histology assess parameter including pigmentation
Immunohistochemical changes in inflammation in all 5 subjects | Visit 2 (Day 28±5) and Visit 5 (Day 112 ±5)
  Histology assess parameter including inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No